CLINICAL TRIAL: NCT02289118
Title: [18F]-T807 PET/CT Imaging of Tau Pathology in Young Onset Focal Dementia
Brief Title: Tau Imaging in Young Onset Dementia
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 820665
Record Dates: First submitted 2014-11-05; First posted 2014-11-13 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer's Disease, Early Onset; Logopenic Progressive Aphasia; Posterior Cortical Atrophy (PCA)
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic Imaging: [18F]T807 imaging tracer.
  Interventions: Drug: [18F]-T807 imaging tracer

INTERVENTIONS:
Drug: [18F]-T807 imaging tracer — Tau Imaging tracer
  Other Names: AV-1451

SUMMARY:
The central goal of this study is to determine and compare the similarities and differences in regional brain uptake of [18F]T807 in patients with typical Alzheimer's Disease (AD), Posterior Cortical Atrophy (PCA), and Logopenic Variant of Primary Progressive Aphasia (lvPPA). The investigators will correlate patterns of [18F]T807 binding with magnetic resonance imaging (MRI)-based regional volumetric and cortical thickness measures. If cerebral spinal fluid (CSF) samples are not available, patients may be asked to get an optional lumbar puncture (LP) for additional comparisons. The investigators will recruit 20 participants, 45-70 years old, with clinical evidence of young onset focal dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be 45 - 70 years of age
2. MMSE > 10 at screening visit.
3. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures. If the patient is unable to provide informed consent, the patient's legal representative may consent on behalf of the patient but the patient will be asked to confirm assent.
4. Participants must be willing and able to comply with scheduled visits and imaging procedures.
5. A brain MRI is required. If a brain MRI has been performed within 6 months of enrollment to this study and of adequate quality that scan may be used for the study analysis, subjects who do not have a brain MRI will undergo a brain MRI either as a part of this study
6. Participants must identify a study partner who is willing to accompany the patient to study visits

Exclusion Criteria:

1. Females who are pregnant or breast feeding at the time of screening scan will not be eligible for this study, urine or serum pregnancy test will be performed in women of child-bearing potential at the time of screening
2. Inability to tolerate or contraindication to imaging procedures (PET/CT or MRI) in the opinion of an investigator or treating physician
3. QTc > 450 msec on screening ECG.
4. Any medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study (e.g. moderate to large stroke or history of moderate or severe traumatic brain injury (TBI)).

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with early onset AD (symptoms preceding age 65)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Determine and compare the similarities and differences in regional brain uptake of [18F]T807 by using standardized uptake value ratio (SUVr) in patients with typical AD, PCA and lvPPA | 2 years
Correlate patterns of [18F]T807 binding based on standardized uptake value ratio (SUVr) with MRI-based regional volumetric (mm3) and cortical thickness (mm) measures | 2 years

SECONDARY OUTCOMES:
Correlate CSF markers of amyloid (Aβ1-42) and/or tau (total tau, phospho-tau) pathology (pg/mL) to uptake of [18F]T807 based on standardized uptake value ratio (SUVr). | 2 years
Correlate [18F]T807 binding based on standardized uptake value ratio (SUVr) with standard cognitive tests. | 2 years
  Neurocognitive test results

CONTACTS AND LOCATIONS:
Overall Officials: David Wolk, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States